CLINICAL TRIAL: NCT06820515
Title: American Thrombosis and Hemostasis Network ATHNdataset Registry
Brief Title: ATHNdataset Registry
Status: Enrolling by invitation | Type: Observational
Sponsor: American Thrombosis and Hemostasis Network (Network)
Responsible Party: Sponsor
Other Study IDs: Pro00082318
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Hemophilia; Thrombosis; Hemophilia A; Hemophilia B; Sickle Cell Disease; Glanzmann Thrombasthenia; Bleeding Disorder; Blood Disorder; Von Willebrand Diseases
Keywords: bleed event; bleed treatments; adverse events; joint bleed; bleeding disorder; bleeding symptoms
MeSH Terms: conditions — Hemophilia A; Thrombosis; Hemophilia B; Anemia, Sickle Cell; Thrombasthenia; Hemostatic Disorders; Hematologic Diseases; von Willebrand Diseases; Hemarthrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Blood Disorders: The ATHNdataset is a large, robust real-world registry that can be queried to produce curated subsets of data to support clinical care, outcomes analysis, safety monitoring, practice of treatment, advocacy, public health reporting, quality improvement projects, and research initiatives. Initiatives relying on the ATHNdataset may focus on gaining a greater understanding of blood disorders, the complications of these disorders, their social and economic costs, and the effectiveness of treatments.
  The population includes all individuals diagnosed with or suspected to have a blood disorder. Participants will contribute data gathered during care encounters with an ATHN Affiliate.

SUMMARY:
The Hemophilia Treatment Center (HTC) where you receive care is working with The American Thrombosis and Hemostasis Network (ATHN) to look at the quality of life of people with blood disorders and problems.

Doctors, scientists, policymakers, and other health care providers need a large amount of information from a lot of people to answer scientific, public health, and policy questions about better ways to treat blood disorders. They will use the information from the ATHNdataset to answer these questions.

DETAILED DESCRIPTION:
Participants who agree to participate will let their health information be included in the ATHNdataset Registry, and the information will be updated regularly to reflect the participant's current health status. This registry includes collecting, storing and managing health information through a secure database. The following health information will be collected:

* Demographics (e.g., age, gender, income, education/occupation)
* The type of blood disorder you have
* Date you were diagnosed, or symptoms began
* Family history of the disorder
* Testing and assessments
* Physical exams
* Height, weight
* Vital signs, including blood pressure and heart rate
* Laboratory tests (results from blood or urine testing, or biological specimens)
* Genetic test results
* Imaging results (X-rays, CT scans, etc.)
* Pharmacokinetic testing results (how drugs are processed in the body)
* Medications used and any problems with use
* Types of bleeds, pain and clotting problems
* Treatments that stop your bleeding or clotting problems from occurring or getting worse
* Surgeries and/or procedures
* Immunizations (vaccines)
* Devices
* Routine care visits and injuries (trauma)
* Other illnesses and diseases you may have
* Allergies
* Patient-reported outcomes (PROs), questionnaires, and surveys
* Payment details for treatment, including insurance companies and health plans

ELIGIBILITY:
Inclusion Criteria:

* Any participant evaluated for or the potential to have a blood disorder who has an encounter with an ATHN Affiliate.
* Participants of any age.
* Participant is able to provide consent or assent; a Legally Authorized Representative (LAR) may provide consent on a participant's behalf if a participant is unable to provide self-consent

Exclusion Criteria:

* Any participant unable to provide consent or assent to participate in the ATHNdataset

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: * Data from participants who have previously provided authorization or consent (according to local requirements) and contributed data to the ATHNdataset will be retained. These participants will be offered a chance to provide updated consent if possible.
  * All future participants from ATHN Affiliates, who meet eligibility criteria and are able to provide consent or assent, will be enrolled prospectively.
  * Participants who have previously contributed data to the ATHNdataset under the terms of an authorization form, an informed consent form, or an assent form will be offered an opportunity to consent.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2024-10-25 (Actual); Primary Completion 2054-10-25 (Estimated); Study Completion 2055-10-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive real-world clinical data registry analysis, research, advocacy, and public health reporting for the blood disorders community | 15 years
  The ATHNdataset Registry objective is to develop a secure, comprehensive registry of real-world clinical data to support standardized comprehensive health information for persons living with blood disorders and public health reporting for the blood disorders community

SECONDARY OUTCOMES:
Contribute to scientific and public health reporting for the blood disorders community | 20 years
  By providing a comprehensive registry for physicians, scientists, policy makers, and other health care stakeholders who require a large pool of participant information to answer questions related to blood disorders treatments

CONTACTS AND LOCATIONS:
Overall Officials: Tammuella Chrisentery-Singleton, M.D., Principal Investigator — American Thrombosis and Hemostasis Network
Locations (1):
- American Thrombosis and Hemostasis Network, Hickory, North Carolina, United States